CLINICAL TRIAL: NCT05927922
Title: Effect of Preoperative Oral Ibuprofen on Anesthetic Efficacy of Inferior Alveolar Nerve Block With Supplemental Buccal and Lingual Infiltrations Using Articaine in Mandibular Molar Teeth With Irreversible Pulpitis: A Randomized Controlled Double-blind Study
Brief Title: Effect of Preoperative Oral Ibuprofen on Anesthetic Efficacy of Inferior Alveolar Nerve Block With Supplemental Buccal and Lingual Infiltrations Using Articaine in Mandibular Molar Teeth With Irreversible Pulpitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abd El hamed, Mohamed Ahmed Abdelhameed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO 3/7/1
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Mandibular Molar Teeth With Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be a double-blinded randomized controlled trial where the patient & operator will not be aware of the intervention used.
  -the treatment groups will be anonymous to the assessing statistician at the end of the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Premedication with 600 mg of Oral Ibuprofen (Experimental): Premedication with 600 mg of Oral Ibuprofen (Abbott, Egypt) will be given 1 hour before IANB.
  Interventions: Drug: Oral Ibuprofen (Abbott, Egypt)
- Placebo will be given 1 hour before inferior alveolar nerve block (Placebo Comparator)
  Interventions: Drug: Oral Ibuprofen (Abbott, Egypt)

INTERVENTIONS:
Drug: Oral Ibuprofen (Abbott, Egypt) — ibuprofen is analegisic drug used to relieve pain

SUMMARY:
Effect of preoperative oral Ibuprofen on anesthetic efficacy of inferior alveolar nerve block with supplemental buccal and lingual infiltrations using articaine in mandibular molar teeth with irreversible pulpitis.

DETAILED DESCRIPTION:
Control group: Placebo will be given 1 hour before IANB. Intervention group: Premedication with 600 mg of Oral Ibuprofen (Abbott, Egypt) will be given 1 hour before IANB.

A sequence of Procedural steps:

1. Clinical and radiographic examination will be done for each tooth.
2. Full medical and dental history will be obtained from all the patients participating in this study, patients will be checked for eligibility and will be informed about the study and sign consent form (Appendix 2) explaining the aim of the trial and the exact steps.
3. Each patient will be given a pain scale chart (Appendix 3) and will be instructed on how to use it. Pre-operative pain level will be recorded.
4. a tooth will be anesthetized using IANB by 3.6 ml of 4 % articaine with 1:100000 adrenaline (Artinibsa, Inibsa Co. for pharmaceuticals & chemical industries, Spain) followed by 0.9mL BI and 0.9 mL LI of 4% articaine with 1:100000 adrenaline (Artinibsa, Inibsa Co. for pharmaceuticals & chemical industries, Spain) using a standard dental aspirating syringe with a 27-G needle. After 15 minutes of the initial IANB, each patient will be asked if his or her lip is numb. If profound lip numbness is not recorded within 15 minutes, the block is considered unsuccessful, and the patients are excluded from the study. If lip numbness is recorded, the patients were further given BI and LI.
5. In the control group: patients will be given a placebo 1 hour before I.A.N.B.
6. In the intervention group: oral administration of 600 mg Ibuprofen (Abbott Pharma, Egypt.) will be given to the patients 1 hour before administration with IANB. After that, same procedures will be followed exactly as the control group.
7. When full lip numbness appears, a sensitivity test for the tooth will be recorded. After 5 minutes from the supplemental injection, the involved teeth will be isolated with a rubber dam and a conventional access opening will be initiated. Patients will be instructed to raise their hand if any pain is felt during any stage of root canal treatment procedure. In case of pain, the procedure will be stopped, and patients will be asked to rate the pain on the VAS.
8. Intraligamentry injection will be given to the patient who recorded Pain intensity greater than will be recorded as well as the step in which the patient felt pain.
9. Root canal treatment procedures will be done as follow:

   * Access cavity will be performed using a round bur and an endo-Z bur (DENTSPLY, Switzerland). The canals will be explored with #10, and #15 K-type hand files (Dentsply Maillefer, Ballaigues, Switzerland) according to the curvature and the initial root canal diameter using a watch-winding motion.
   * The working length (WL) will be established using a Root ZX mini apex locator (J Morita Corp, Kyoto, Japan), and will be confirmed radiographically.
   * The root canals will be thoroughly irrigated using 3ml syringe of 2.5% sodium hypochlorite (Clorox, 10th of Ramadan, Egypt) with irrigant flow rates ranging from 0.03 ml/sec to 1.27 ml/sec. after each instrument. A side vented needle (Diadent, Chungcheongbuk-do, Korea) will be used shorter than the working length by 1mm to control the possibility of irrigant apical extrusion.22
   * Cleaning and shaping of all root canals will be carried out using M PRO (IMD, Shanghai, China) rotary files for both groups in a continuous rotary brushing motion, following the manufacturer's instructions. A gear reduction torque-controlled X-smart motor (Dentsply Maillefer, Maillefer, USA) will be used. For the first two-thirds of the working length, file (18/.09) served as an orifice opener in a continuous rotation motion with 500 rpm speed and 3 Ncm torque. Following that, (20/.04) and (25/.06) will be used respectively for the remaining working length at 500 rpm and 1.5 Ncm of torque. The files will be used in & out motions of 3mm stroke length each time until reaching the working length. After using each file, the canal will be recapitulated and irrigated using 2 ml NaOCl. The apical portion of distal canals will be manually enlarged to size #35k file.
   * Master cones selection will be done and confirmed radiography.
   * Root canal irrigation will be done using saline followed by 3 ml 17% EDTA (META, Chungbuk, ROK) for 1 min to remove the smear layer.
   * Canals will be dried using sterile paper points (Meta Biomed Co. Ltd, Korea), and then will be obturated using a resin-based sealer ADSEAL (META BIOMED Co., LTD., Chungbuuk, Korea) with the lateral compaction technique.
10. The access cavity will then be closed with an intermediate restorative material (MD Temp temporary filling) to ensure a good coronal seal. A post-operative radiograph will be obtained.
11. Adverse effects such as pain during and after injection will be recorded for each patient.
12. Post-operative instructions will be given to all patients. • The patient will be asked to rate their post-operative pain level 6, 12, 24, and 48 hours postoperatively according to the given instructions and will be asked to return for a follow-up after 2 days to hand the pain scale chart (HP VAS scores)

Outcome:

Primary outcome:

The success rate of local anesthesia through measuring pain during root canal treatment using HP

VAS. It is a line numbered from 0-170mm, where pain levels are categorized as follows:

* "0" = no pain
* 1-54mm = faint, weak, or mild pain
* 55-114mm = moderate pain
* 114-170mm = strong, intense, or severe pain, "170mm" is the most intense pain. where success is defined as no or mild pain (0-54mm) throughout the procedure.

Secondary outcome:

Degree of postoperative pain using a modified visual analog scale. It is a line numbered from 0-10, where pain levels are categorized as follows:

* "0" = no pain
* 1-54mm = faint, weak, or mild pain
* 55-114mm = moderate pain
* 114-170mm = strong, intense, or severe pain, "170mm" is the most intense pain.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with age between 18-50 years.
2. Systemically healthy patients (ASA I or II).
3. patient's signs and symptoms give diagnosis of symptomatic irreversible pulpitis in mandibular molar teeth including: i. Presence of sharp pain upon thermal stimulus, lingering pain (often 30 seconds or longer after stimulus removal), spontaneity (unprovoked pain) and referred pain (According to American Association of Endodontics, 2013). According to Azim et al (2022), a clinical diagnosis for symptomatic irreversible pulpitis based on subjective (lingering pain to thermal changes for extended period).

ii. Pre-operative sharp pain marked on VAS scale by reading not less than 6. iii. exaggerated response with continuous lingering pain to cold pulp tester using ethyl chloride spray (Walter Ritter Gmbh +Co.-pharmaceutical - Germany. The Egyptian pharmaceutical trading company) and electric pulp tester (Denjoy dental CO., LTD.Changsha.P.R China).

iv. Normal periapical radiographic appearance or slight widening of the periodontal ligament space.

v.Presence of objective findings such as caries or fracture, deep restorations. vi. No pain on percussion.

-

Exclusion Criteria:

1. Allergy to articaine or Ibuprofen
2. History of intolerance to NSAIDs.
3. Patients who have taken analgesics or anti-inflammatory drugs 12 hours before treatment.
4. Patients with two or more adjacent teeth requiring endodontic treatment.
5. Pregnant or nursing females.
6. Teeth that have periodontal affection (with a pocket depth greater than 5mm, associated with swelling or fistulous tract, or greater than grade I mobility)
7. Non-restorable teeth.
8. Teeth fracture and resorption.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Success rate of local anesthesia | During access cavity preparation and cleaning and shaping procedures of root canal treatment.
  Success rate of local anesthesia through measuring pain during root canal treatment using HP
  VAS. It is a line numbered from 0-170mm, where pain levels are categorized as follows:
  * "0" = no pain
  * 1-54mm = faint, weak or mild pain
  * 55-114mm = moderate pain
  * 114-170mm = strong, intense or severe pain, "170mm" being the most intense pain conceivable.
  where success is defined as no or mild pain (0-54mm) throughout the procedure

SECONDARY OUTCOMES:
Degree of post-operative pain | 6, 12, 24 and 48 hours post-operatively.
  Degree of post-operative pain using modified visual analogue scale. It is a line numbered from 0-10, where pain levels are categorized as follows:
  * "0" = no pain
  * 1-54mm = faint, weak or mild pain
  * 55-114mm = moderate pain
  * 114-170mm = strong, intense or severe pain, "170mm" being the most intense pain conceivable

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes